CLINICAL TRIAL: NCT00882427
Title: Single-center, Open Study on the Performance of the Software eMPC Algorithm Used for Blood Glucose Control Over an Extended Glucose Control Range (4.4 to 8.3 mmol/L) for a Maximum of 48 Hours in Postoperative Cardiac Surgery Patients in the Intensive Care Unit
Brief Title: Blood Glucose Control Over an Extended Glucose Control Range in Postoperative Cardiac Surgery Patients in the Intensive Care Unit
Acronym: Aldea_02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Dr. Norman Kachel, B. Braun Melsungen AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC-G-H-0807
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Critical Illness
Keywords: algorithm; tight glycemic control; glucose control; intensive care; insulin; ICU
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eMPC (Experimental): improved model predictive control algorithm (eMPC) for glycaemic control in ICU patients
  Interventions: Other: enhanced model predictive control algorithm (eMPC)

INTERVENTIONS:
Other: enhanced model predictive control algorithm (eMPC) — eMPC (software on a bedside computer) advised insulin titration to establish tight glycaemic control

SUMMARY:
Hyperglycaemia is commonly found in critically ill patients. Clinical studies demonstrated that tight blood glucose control in medical and surgical ICU patients results in a significant better outcome for the patients. Based on this emerging clinical evidence, there are increasing efforts worldwide to maintain strict glycaemic control in critically ill patients. However, achieving this goal requires extensive nursing efforts, including frequent bedside glucose monitoring and the implementation of complex intensive insulin infusion protocols. A fully automated algorithm may help to overcome some of these limitations by excluding intuitive interventions and integrating relevant clinical data in the decision-making process. This study will investigate the performance of an eMPC algorithm adjusted to target the range 4.4 - 8.3 mmol/L in line with the Surviving Sepsis guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years of age
* Admitted following cardiac surgery
* Stay in the ICU expected to be > 20h
* Blood glucose > 6.7 mmol/l within 4 hours of admission to intensive care or patient already receiving insulin treatment

Exclusion Criteria:

* Patients with hyperglycaemic crisis/ketoacidosis due to insulin deficiency.
* Known or suspected allergy to insulin
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient (i.e. liver failure, other fatal organ failures)
* Patients participating in another study
* Moribund patients likely to die within 24 hours
* Patients after organ transplantation within the last three months
* Patients under high dose cortisol treatment (cortisol > 1000 mg/day or equivalent doses of hydrocortisol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
percentage of time within the predefined glucose target range of 80-150 mg/dL | from start of treatment to the last glucose measurement under treatment

SECONDARY OUTCOMES:
Hypoglycemias | from start of treatment to the last glucose measurement under treatment
Usability parameters like convenience of alarming function; workload; blood sampling frequency | from start of treatment to the last glucose measurement under treatment
Concomitant medication including insulin infusion rate, parenteral/enteral nutrition | from start of treatment to the last glucose measurement under treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Cordingley, Dr., Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital and Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Cordingley JJ, Vlasselaers D, Dormand NC, Wouters PJ, Squire SD, Chassin LJ, Wilinska ME, Morgan CJ, Hovorka R, Van den Berghe G. Intensive insulin therapy: enhanced Model Predictive Control algorithm versus standard care. Intensive Care Med. 2009 Jan;35(1):123-8. doi: 10.1007/s00134-008-1236-z. Epub 2008 Jul 26. PMID 18661120